CLINICAL TRIAL: NCT05123768
Title: Evaluation of Genetic Etiology in Patients With Cerebral Palsy
Brief Title: Genetic Etiology in Patients With Cerebral Palsy
Acronym: GenCP
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Damjan Osredkar, Associate Professor Damjan Osredkar, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: 0120-142/2021/2
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Palsy; Genetic Disease; Developmental Delay; Metabolism, Inborn Errors
Keywords: Cerebral palsy; Genetic disease; Neurodevelopmental disorder; Inborn errors of metabolism; Spasticity; Dystonia; Ataxia; Next generation sequencing; Aromatic l-amino acid decarboxylase deficiency
MeSH Terms: conditions — Cerebral Palsy; Genetic Diseases, Inborn; Learning Disabilities; Metabolism, Inborn Errors; Neurodevelopmental Disorders; Muscle Spasticity; Dystonia; Ataxia; Aromatic amino acid decarboxylase deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — DNA will be extracted from whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cerebral palsy: In Slovenia, all children with cerebral palsy born in 1996 or later are included in the Slovenian National Registry of Cerebral Palsy. All patients from the Registry will be invited to participate in the study.
  Interventions: Diagnostic Test: NGS

INTERVENTIONS:
Diagnostic Test: NGS — A genetic panel of more than 100 genes, associated with CP spectrum disorders, will be assessed using NGS
  Other Names: Next gen sequencing

SUMMARY:
Cerebral palsy (CP) is a permanent disorder of movement or posture due to non-progressive impairments of the developing brain. Current estimates indicate that as many as 30% of CP cases may be genetic in nature. In our study, the investigators will re-examine the data of children with CP, who are registered in the Slovenian National Registry of Cerebral Palsy. All children will be invited to the University Children's Hospital, University Medical Centre Ljubljana, where they will be re-examined by a neurologist. Blood for genetic testing will be taken. In the case of confirmed genetic ethiology of CP, the search for specific therapy will be possible.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a permanent disorder of movement or posture due to non-progressive impairments of the developing brain. In children, CP is the most common cause of motor impairment, which is often accompanied by other disorders such as epilepsy, mental retardation, speech and language disorders, eating disorders, visual and hearing disorders, and behavioral disorders. Approximately 1 child in every 500 live births is diagnosed with cerebral palsy.

The causes of CP are usually related to inadequate blood flow and oxygen supply to the baby's central nervous system during pregnancy or birth, complications of premature birth, and other complications in the neonatal period such as respiratory distress, infections, or jaundice. It is estimated that in up to one third of children with CP the cause is unexplained. The cause of CP in these children may also be rare genetic diseases. For some of these diseases a targeted treatment is available.

In Slovenia, all children with CP, born since 1996, are included in the Slovenian National Registry of Cerebral Palsy (SRCP), which is part of the European registry - Surveillance of Cerebral Palsy in Europe (SCPE). Children are entered into the register at University Children's Hospital, University Medical Centre Ljubljana at the age of 5, after prior parental consent, otherwise anonymously.

In our study, the investigators will re-examine the data of children with CP, who are registered in the SRCP. All children will be invited to the University Children's Hospital, University Medical Centre Ljubljana, where they will be re-examined by a neurologist. With the consent of the patient or his/her parent/guardian, blood for genetic test will be taken. Utilising next gen sequencing (NGS), a gene panel of more than 100 genes associated with the CP spectrum disorders will be performed. In the case of confirmed genetic ethiology of CP, the search for specific therapy will be possible.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy who are included in the Slovenian National Register of Cerebral Palsy (SRCP)
* Patients whose parents/caregivers were informed about the aims of the study and have signed the Informed consent form.

Exclusion Criteria:

* Patients who are not diagnosed with cerebral palsy
* Patients whose caregivers have not signed the Informed consent form.

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will enroll and collect data from children with cerebral palsy of any grade (I-V) who are included in the Slovenian National Register of Cerebral Palsy (SRCP) and whose parents/caregivers were informed about the aims of the study and have signed the Informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Identification of genetic etiology | 2-3 months after collection of DNA samples
  Next gen sequencing (NGS) will be performed and a panel of over 100 genes will be evaluated for identification of potential genetic etiology.

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No